CLINICAL TRIAL: NCT00964886
Title: Efficacy of Antidepressants in Chronic Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NURA-019-09S
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Back Pain
Keywords: chronic pain; back pain; antidepressants
MeSH Terms: conditions — Back Pain; Chronic Pain | interventions — Cognitive Behavioral Therapy; Desipramine; Clomipramine; Benztropine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental): desipramine hydrochloride
  Interventions: Drug: desipramine hydrochloride
- Arm 2 (Experimental): cognitive behavioral therapy
  Interventions: Behavioral: cognitive behavioral therapy
- Arm 3 (Experimental): desipramine hydrochloride and cognitive behavioral therapy
  Interventions: Drug: desipramine hydrochloride; Behavioral: cognitive behavioral therapy
- Arm 4 (Placebo Comparator): anticholinergic medication; active placebo
  Interventions: Drug: benztropine mesylate 0.125 mg daily

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — cognitive behavioral therapy, a type of psychotherapy oriented towards restoring function and reducing impact of pain on everyday life
  Arms: Arm 2
Drug: desipramine hydrochloride — desipramine hydrochloride, with dose targeted to achieve a serum concentration of 5-60ng/ml
  Other Names: Anafranil
  Arms: Arm 3
Behavioral: cognitive behavioral therapy — cognitive behavioral therapy, a type of psychotherapy oriented towards restoring function and reducing impact of pain on everyday life
  Arms: Arm 3
Drug: benztropine mesylate 0.125 mg daily — benztropine mesylate is a placebo, some of whose side effects mimic those of experimental intervention, desipramine hydrochloride
  Other Names: Cogentin
  Arms: Arm 4
Drug: desipramine hydrochloride — desipramine hydrochloride, with dose targeted to achieve a serum concentration of 5-60ng/ml
  Other Names: Anafranil
  Arms: Arm 1

SUMMARY:
This 12 week placebo controlled clinical trial tests the individual and combined effects of an antidepressant medication and cognitive behavioral therapy for chronic back pain.

DETAILED DESCRIPTION:
This is a 4 arm 12 week randomized clinical trial comparing the efficacy of 1) low concentration desipramine (< 60 ng/ml); 2) cognitive behavioral therapy; 3) low concentration desipramine + cognitive behavioral therapy; and 4) placebo medication (benzotropine mesylate).

ELIGIBILITY:
Inclusion Criteria:

* Chronic back pain (daily pain for > 6 months)

Exclusion Criteria:

* Major medical conditions which might contraindicate antidepressant treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph H Atkinson, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Available in SPSS format from the investigators.

REFERENCES:
- [Derived] Gould HM, Atkinson JH, Chircop-Rollick T, D'Andrea J, Garfin S, Patel SM, Funk SD, Capparelli EV, Penzien DB, Wallace M, Weickgenanta AL, Slater M, Rutledge T. A randomized placebo-controlled trial of desipramine, cognitive behavioral therapy, and active placebo therapy for low back pain. Pain. 2020 Jun;161(6):1341-1349. doi: 10.1097/j.pain.0000000000001834. PMID 32068667

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Started | 38 | 34 | 37 | 33
Completed | 27 | 27 | 21 | 24
Not Completed | 11 | 7 | 16 | 9
Not completed — Lost to Follow-up | 2 | 2 | 6 | 4
Not completed — Withdrawal by Subject | 6 | 2 | 5 | 3
Not completed — Adverse Event | 3 | 1 | 5 | 2
Not completed — Protocol Violation | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic characteristics of participants randomized at baseline to one of the four study arms (selected information on three participants missing)
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 37 | 33 | 37 | 32 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (11.7) | 57.8 (9.2) | 51.5 (13.7) | 57.9 (10.9) | 55.8 (11.7)
Gender [Count of Participants; unit: Participants] — Population: Gender data missing on one participant.
  Participants
    number analyzed (Participants) | 37 | 33 | 37 | 31 | 138
    Female | 5 | 4 | 3 | 3 | 15
    Male | 32 | 29 | 34 | 28 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 5 | 4 | 25
  Not Hispanic or Latino | 29 | 22 | 28 | 24 | 103
  Unknown or Not Reported | 2 | 1 | 4 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data missing on one participant.
  Participants
    number analyzed (Participants) | 37 | 32 | 37 | 32 | 138
    American Indian or Alaska Native | 0 | 2 | 1 | 0 | 3
    Asian | 1 | 1 | 2 | 1 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2
    Black or African American | 6 | 6 | 4 | 5 | 21
    White | 25 | 18 | 21 | 20 | 84
    More than one race | 4 | 2 | 7 | 3 | 16
    Unknown or Not Reported | 1 | 3 | 1 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 37 | 33 | 37 | 32 | 139
Pain Intensity and Back Pain Disability [Mean (Standard Deviation); unit: units on a scale] — The DDS is self-report measure of "current" pain intensity on a 20 point scale relative to 12 adjectival descriptor words which serve as anchors (eg, greater or less than "faint," "moderate," "strong"). Scores range from 0 to 20 with higher scores indicating higher pain intensity.
  The Roland and Morris questionnaire is a 24-item checklist asking patients whether or not back pain limits activities they normally do (eg, "I stay at home most of the time because of my back"). Scores range from 0 to 24, with higher scores indicating greater disability in everyday function due to back pain
  units on a scale
    Pain Intensity (Descriptor Differential Scale) | 9.9 (4.9) | 11.9 (4.3) | 11.9 (5.1) | 12.1 (4.6) | 11.4 (4.0)
    Back Pain Disability (Roland and Morris) | 8.7 (5.4) | 13.0 (4.3) | 11.7 (5.4) | 12.6 (3.8) | 11.8 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Intent-toTreat Analysis of Descriptor Differential Scale (DDS) of Pain Intensity
Description: The DDS is self-report measure of "current" pain intensity of chronic back pain. Participants rate pain on a 20 point scale as being greater or less intense relative to 12 adjectival descriptor words which serve as anchors (eg, greater or less than "faint," "moderate," "strong"). Scores range from 0 to 20 with higher scores indicating higher pain intensity. The analysis evaluated the 'as randomized' sample at 12 weeks after baseline or last observation carried forward, after co-varying for baseline (pre-treatment) values.
Time Frame: 12 weeks after baseline (or last observation carried forward)
Population: We conducted an intent-to-treat analysis of all randomized participants assigned to desipramine or to active drug placebo (benztropine) comparing mean DDS pain intensity at Week 12 (or the last observation carried forward) adjusted for mean baseline score.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Arm 1 + Arm 3: Factor desipramine hydrochloride
  desipramine hydrochloride: desipramine hydrochloride, with dose targeted to achieve a serum concentration of 5-60ng/ml
- Arm 2 + Arm 4: Factor anticholinergic medication; active placebo
  benztropine mesylate 0.125 mg daily: benztropine mesylate is a placebo, some of whose side effects mimic those of experimental intervention, desipramine hydrochloride
Arm/Group | Arm 1 + Arm 3 | Arm 2 + Arm 4
Number analyzed (Participants) | 75 | 67
units on a scale | 8.3 (0.5) | 8.1 (0.6)
Statistical Analysis 1: Comparison: Arm 1 + Arm 3 vs Arm 2 + Arm 4; In an intent-to-treat analysis of all randomized participants assigned to experimental drug (desipramine) or active placebo (benztropine) an analysis of variance compared mean Descriptor Differential Scale scores at 12 weeks (or last observation carried forward) adjusted fro mean baseline score ( = ); Test type: Superiority or Other; p = 0.7, ANCOVA

2. Secondary Outcome: Roland and Morris Disability Questionnaire
Description: This questionnaire measures disability in everyday function due to back pain. It is a 24-item checklist asking patients to endorse whether or not back pain limits activities they normally do (eg, "I stay at home most of the time because of my back"). Scores range from 0 to 24, with higher scores indicating greater disability in everyday function due to back pain. The analysis evaluated the 'as randomized' sample at 12 weeks after baseline, after co-varying for baseline (pre-treatment) values.
Time Frame: 12 weeks after baseline (or last observation carried forward)
Population: All participants assigned at baseline to receive desipramine hydrochloride or benztropine mesylate (drug effect). This is an 'as randomized' Intent-to-Treat analysis. Values are mean scores at Week 12 (or last observation carried forward). Means are adjusted for baseline Roland and Morris scores
Measure: Mean (Standard Error); unit: Units on a scale.
Groups:
- Arm 1 + Arm 3: Factor all participants assigned at baseline to receive desipramine hydrochloride
- Arm 2 + Arm 4: Factor all participants assigned at baseline to receive benztropine mesylate (active placebo)
Arm/Group | Arm 1 + Arm 3 | Arm 2 + Arm 4
Number analyzed (Participants) | 75 | 67
Units on a scale. | 8.7 (0.5) | 8.9 (0.5)
Statistical Analysis 1: Comparison: Arm 1 + Arm 3 vs Arm 2 + Arm 4; In the intent-to-treat sample of all randomized participants assigned to experimental drug (desipramine) or active placebo (benztropine) an analysis of variance (ANOVA) compared mean Roland and Morris scores at 12 weeks adjusted for mean baseline scores; Test type: Superiority or Other; p = 0.84, ANCOVA; Means are adjusted for baseline Roland and Morris scores

3. Primary Outcome: Intent-toTreat Analysis of Descriptor Differential Scale (DDS) of Pain Intensity
Description: as for outcome 1
Time Frame: 12 weeks after baseline (or last observation carried forward)
Population: We conducted an intent-to-treat analysis of all randomized participants assigned to cognitive behavioral therapy to or no behavior therapy comparing mean DDS pain intensity at Week 12 (or the last observation carried forward) adjusted for mean baseline score.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Arm 2 + Arm 3: Factor cognitive behavioral therapy
  cognitive behavioral therapy: cognitive behavioral therapy, a type of psychotherapy oriented towards restoring function and reducing impact of pain on everyday life
- Arm 1 + Arm 4: Factor no cognitive behavioral therapy
Arm/Group | Arm 2 + Arm 3 | Arm 1 + Arm 4
Number analyzed (Participants) | 71 | 71
units on a scale | 8.0 (0.6) | 8.4 (0.6)
Statistical Analysis 1: Comparison: Arm 2 + Arm 3 vs Arm 1 + Arm 4; Test type: Superiority or Other; p = 0.6, ANCOVA

4. Secondary Outcome: Roland and Morris Disability Questionnaire
Description: as for outcome 2
Time Frame: 12 weeks after baseline (or last observation carried forward)
Population: All participants assigned at baseline to receive cognitive behavioral therapy or to no cognitive behavioral therapy (behavioral effect). This is an 'as randomized' Intent-to-Treat analysis. Values are mean scores at Week 12 (or last observation carried forward). Means are adjusted for baseline Roland and Morris scores
Measure: Mean (Standard Error); unit: Units on a scale.
Groups:
- Arm 2 + Arm 3: Factor all participants assigned at baseline to receive cognitive behavioral therapy
- Arm 1 + Arm 4: Factor all participants assigned at baseline not to receive cognitive behavioral therapy
Arm/Group | Arm 2 + Arm 3 | Arm 1 + Arm 4
Number analyzed (Participants) | 71 | 71
Units on a scale. | 8.7 (0.5) | 8.9 (0.5)
Statistical Analysis 1: Comparison: Arm 2 + Arm 3 vs Arm 1 + Arm 4; This analysis compares outcomes for participants assigned at baseline to receive cognitive behavioral therapy or not to receive cognitive behavioral therapy (behavioral effect); Test type: Superiority or Other; p = 0.8, ANCOVA

ADVERSE EVENTS:
Time Frame: Report of side effects experienced within the past 3 days by participants completing the Week 12 visit.
Description: Non-serious adverse advents were monitored for 70 participants.
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Serious Adverse Events (participants affected / at risk) | 1/38 | 0/34 | 1/37 | 0/33
Other Adverse Events (participants affected / at risk) | 12/17 | 8/20 | 7/16 | 6/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=38) | Arm 2 (N=34) | Arm 3 (N=37) | Arm 4 (N=33)
urosepsis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalized 2 days after starting study drug (desipramine) for urinary tract infection.
fall (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Fell off bed while attempting to swat an insect on ceiling.Reported to emergency department for treatment of laceration of scalp. After suturing he converted from regular sinus rhythm to atrial fibrillation. Was admitted for cardioversion.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=17) | Arm 2 (N=20) | Arm 3 (N=16) | Arm 4 (N=17)
dry mouth (Gastrointestinal disorders) | 5 (5) | 3 (3) | 4 (4) | 1 (1)
difficulty urinating (Renal and urinary disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 1
erectile dysfunction (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
accomodation disturbance (Eye disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
decreased libido (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
increased dreaming (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
sedation (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
increased sleep duration (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
ejaculatory dysfunction (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
orgasm dysfunction (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
asthenia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
diaphoresis (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
muscle rigidity (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
hyperkinesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
dystonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
gynecomastia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
insomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
nausea (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
photosensitivity (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
weight gain (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Failure to attain recruitment goals and attrition resulted in lack of power to detect an effect. A strong active placebo control condition (benztropine) and frequent follow up visits may have led to improvement in all groups over time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes